CLINICAL TRIAL: NCT00709839
Title: Rapid Effects of Hydrocortisone on Glucose-induced Insulin Secretion in Healthy Humans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Anton Luger, Department of Medicine III, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FSIGT_Hydrocortisone_01
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: glucocorticoid; hydrocortisone; carbohydrate metabolism; appetite-regulatory hormones
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hydrocortisone — 0.6 mg/kg body weight, intravenous bolus given at time-point minus 4'
Drug: Glucose 33% — 1ml/kg body weight, intravenous bolus given at time-point 0'

SUMMARY:
The purpose of this study is to investigate the effect of hydrocortisone on glucose-induced insulin secretion and sensitivity, by means of an intravenous glucose tolerance test with frequent sampling (FSIGT) followed by minimal model analysis. In a randomized single-blind cross-over design, the subjects will receive either hydrocortisone or placebo 4 minutes before an intravenous glucose load.

DETAILED DESCRIPTION:
Glucocorticoids (mainly cortisol in men and corticosterone in rodents) are secreted in the adrenal cortex under the control of the hypothalamic-pituitary-adrenal (HPA) axis. They are known for and named after their combined actions on glucose metabolism: suppression of insulin secretion, inhibition of glucose uptake in peripheral tissues, and promotion of gluconeogenesis in the liver. As a result, glucose intolerance accompanies syndromes of cortisol excess, while recurrent hypoglycemia, especially in response to stress, is a typical feature of isolated familial glucocorticoid deficiency. Almost any acute severe challenge to homeostasis or stress will activate the hypothalamic-pituitary-adrenal (HPA) axis and cause a rise in plasma glucocorticoid levels, which is essential for survival. Thanks to their immunosuppressive and antiinflammatory actions, glucocorticoids are widely-used therapeuticals with important adverse effects.

The need to optimize the benefit-risk ratio of glucocorticoid therapy has lead to a recent focus of research in the pathways mediating their effects. Glucocorticoids act rapidly and within minutes, exerting effects which contradict the classical genomic signalling pathway. Little is known on the clinical rapid effects of glucocorticoids on carbohydrate metabolism. Corticosterone acutely lowers insulin plasma concentrations and their response to hyperglycemia in rodents in vivo. Intraperitoneally administered hydrocortisone suppresses the insulin levels stimulated by intravenous glucose in mice. Although subject to numerous studies, the metabolic effects of glucocorticoids have been generally tested after giving dexamethasone for a few days.

To our knowledge, there are no data on rapid effects of glucocorticoids on insulin secretion and sensitivity in humans. Despite the increased interest in rapid effects of steroids in the last decade, the immediate effects of glucocorticoids on carbohydrate metabolism have not yet been studied. This question is not easy to address in vivo because of the multiple (also compensatory) influences that can impact the endocrine pancreas. Therefore, we propose to use a rapid approach, studying the effect of a bolus of hydrocortisone on the response to an intravenous glucose tolerance test with frequent sampling (FSIGT).

The FSIGT consists in giving intravenously a glucose bolus and taking frequently blood samples afterwards for determining glucose, insulin and C-peptide. The glucose and insulin data analysed with the minimal model technique allow the calculation of the acute insulin response, glucose effectiveness and the insulin sensitivity index. The data on C-peptide will be used to evaluate the beta cell function.

The effects of Hydrocortisone on glucose-induced insulin secretion and sensitivity will be investigated by means of an FSIGT followed by minimal model analysis. The subjects will receive in a randomized single-blind cross-over design:

1. 0.6 mg/kg body wt Hydrocortisone + 330 mg/kg body wt glucose
2. Placebo + 330 mg/kg body wt glucose

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* No concomitant medication
* BMI < 25 kg/m2
* Age: 18-60 years old

Exclusion Criteria:

* Impaired glucose tolerance or diabetes mellitus
* Hyperthyroidism, hypothyroidism
* Hepatic, renal or cardiovascular diseases
* Malignancies
* History of medical therapy within 3 weeks prior to enrolment into the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Plasma insulin, glucose and C-peptide | Minutes: -10, -5, 0, 3, 4, 5, 6, 8, 10, 15, 20, 30, 40, 60, 80, 100, 120, 150, 180

SECONDARY OUTCOMES:
Plasma levels of appetite-regulatory hormones: ghrelin, PYY and nesfatin-1. | Minutes: -10, 0, 30, 60, 120, 180

CONTACTS AND LOCATIONS:
Overall Officials: Anton Luger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Division of Endocrinology and Metabolism, Department of Medicine III, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Result] Vila G, Krebs M, Riedl M, Baumgartner-Parzer SM, Clodi M, Maier C, Pacini G, Luger A. Acute effects of hydrocortisone on the metabolic response to a glucose load: increase in the first-phase insulin secretion. Eur J Endocrinol. 2010 Aug;163(2):225-31. doi: 10.1530/EJE-10-0282. Epub 2010 May 18. PMID 20484150